CLINICAL TRIAL: NCT06599970
Title: Improving Disease Prevention Strategies of Epidemic Spread by Integrating Socio-spatial Characterization of Human Mobility, Environmental Typology and Mathematical Modelling in an Urban System of Cuba
Brief Title: Improving Disease Prevention Strategies by Integrating Socio-spatial Characterization of Human Mobility
Acronym: DI-MOB
Status: Recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Cienfuegos Provincial Ministry of Health, Cuba (Unknown); University Ghent (Other); Institute Pedro Kouri, Ministry of Public Health (Cuba) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 756227
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Dengue; Arbovirus Infections; Epidemic Disease; Behavior, Health
Keywords: human mobility; transmission modelling; socio-spatial characterization
MeSH Terms: conditions — Dengue; Arbovirus Infections; Health Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — This is an observational study. No experimental interventions included. The mobility of people will be studied.

SUMMARY:
In contrast to the trend expected based on existing prediction models, dengue incidence was historically low during the pandemic mobility restrictions of 2020-2021 in most dengue endemic countries. This highlights that current transmission models do not correctly take human mobility into account. Within a pilot-study in Cienfuegos, South-Central Cuba, we will characterise the epidemiological spread and distribution of dengue outbreaks (2012-2025) in districts repeatedly involved in previous dengue outbreaks as initiating, case-concentrating or transmission sustaining areas. This will be linked with fine-grained mobility data and socio-spatial characterizations of commuting flows and population hubs where people are concentrated during day-time (time when transmission happens). This information, together with entomological and environmental risk-data, will be used to i) improve the accuracy of mathematical dengue models, ii) better understand the transmission process and iii) inform and improve the design of disease control strategies. The project will contribute to much-needed evidence-based guidance for public health actors on improved prevention strategies of epidemics dispersion and where and when to implement control measures.

DETAILED DESCRIPTION:
Using epidemiological data and human mobility data, integrated with other multiple-sourced data, this study examines the interplay between disease spread and intra-city mobility (within a city).

The study is ambi-spective, using retro- and prospective routine surveillance data (2012-2025) on dengue cases and Aedes entomological data, to describe the fine-scale spatio-temporal characterization of dengue transmission in Cienfuegos municipality.

To characterise human mobility within the municipality of Cienfuegos, information related to recurrent and seasonal movements will be collected. Several types of data will be triangulated to obtain a comprehensive understanding of the population's mobility (matrix of human mobility). In this way, six prospective data collection activities are planned:

1. Mobility survey: The conduct of a mobility survey with adults. The purpose of this survey is to gather prospective information regarding recurrent mobility, and retrospective information about seasonal mobility. Study subjects include adults, elderly, and indirectly, young children through the specific inclusion of young mothers.
2. Student survey: Questionnaire about mobility of a sample of students in pre-university and university on recurrent and seasonal mobility.
3. School registers: Consultation of school registers to capture information on school-related recurrent mobility of children of school-going age.
4. Vacation stories: Within a two-weeks time after the holidays, teachers are always doing a 'vacation story exercise' within their class. We will ask the teachers of selected classes in the sentinel schools to group this information on the number of children travelling outside the Cienfuegos municipality during holidays (seasonal mobility).
5. Workplace register: Consultation of workplace registers to capture information on work-related recurrent mobility of adults.
6. Call Detail Records: Anonymized and grouped information about house-work/school locations of cell phone users obtained from cell phone company (recurrent movement).

In a third step, the above information will be brought into a mathematical model, explaining mobility within transmission dynamics, which will be validated in a prospective way allowing to identify shortcomings and adjust the model where needed.

In a last step, the various types of collected data will be assembled and discussed together for the elaboration of potential dengue (and integrated) control strategies and presented for validation with local stakeholders.

ELIGIBILITY:
For the prospective data collection - mobility survey:

Inclusion Criteria:

* Being a resident of the sentinel Popular Council/consultorio
* Being >= 19 years of age
* Being willing and able to provide written informed consent

Exclusion Criteria:

* being below 19 or above 75 years old

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Research will take place in Cienfuegos municipality, Cuba, with a population of 178 776 inhabitants. For the epidemiological and entomological data, routine surveillance info will be used, which covers the entire municipality.
  For mobility patterns characterisation, for example the mobility survey: we selected (based on epidemiological patterns) 5 sentinel Popular Councils. Within each, 4 consultorios and their area of coverage were selected. In the consultorium exists a health registry, a list of all persons in the consultorium catchment area. Participants will be selected from the health registry by a random process using the RANDBETWEEN function in Microsoft Excel, within a range of 1 to upper limit equal to the total number of patients in the registry.
Sampling Method: Probability Sample
Enrollment: 810 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
dengue incidence | 2012-2025
  multilevel spatio-temporal characterization of dengue transmission dynamics, focussing on transmission propagation heterogeneity in time and space
human mobility | 2024-2026
  origen-destination matrices will be built, based on information collected in mobility survey, school and workplace registries, vacation stories, phone data, student survey and in-depth interviews

SECONDARY OUTCOMES:
entomological risks for dengue transmission | 2012-2025
  entomological indicators (monthly data collection of immature stages 2012-2025; monthly surveys of adult stages Aedes mosquitoes 2024-2025)
climate | 2012-2026
  temperature (° degrees celsius, daily minimum, daily maximum, weekly average) and rainfall (mm/day)
Mathematical transmission model | 2024-2026
  Stochastic mobility-driven spatially explicit DENV model based on the two primary outcomes of this study
socio-spatial characterisation of public spaces | 2024-2026
  hourly population densities (number of persons present for more than 5 minutes present) in different rooms/areas of densely frequented public spaces (schools, markets, factories)

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Vanlerberghe, Study Director — Institute of Tropical Medicine
Locations (1):
- Instituto de Medicina Tropical Pedro Kouri, Havana, La Habana, Cuba